CLINICAL TRIAL: NCT01238666
Title: Feasibility of a Minimally Invasive Image-Guided Surgery System for Hepatic Ablation Procedures
Brief Title: Evaluation of a Minimally Invasive Image-Guided Surgery System for Hepatic Ablation Procedures
Status: Completed | Type: Observational
Sponsor: Pathfinder Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: PTI-LC-2010-01
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Liver Cancer
Keywords: liver; cancer; tumor; ablation; Pathfinder
MeSH Terms: conditions — Liver Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study was designed in two phases: Phase I is designed to confirm that the surgeon is able to perform accurate liver surface registration including standard liver features used as landmarks during a scheduled laparoscopic liver ablation procedure and acquires a level of comfort with the procedure.

The surface of the liver will be manually swabbed with the study tracked laparoscopic probe with landmarks noted during data collection. After registration of the liver is obtained, the registration points obtained during this procedure will be evaluated by the surgeon by moving the tracked laparoscopic probe over the liver surface and evaluating the location of the tracked laparoscopic probe displayed on the guidance system three dimensional (3D) image. The surgeon will accept or reject the registration accuracy.

The hypothesis is that the surgeon will be able to successfully acquire liver surface registrations with a small learning curve for technique and will be able to proceed to Phase II of the study.

Phase II contains the registration process included above but adds the additional process of tracking the ablation probe used to perform tumor ablation by attaching the Pathfinder Multi-Tool adaptor and collecting data showing the location of the ablation probe as tracked and displayed on the Pathfinder three dimensional (3D) image.

The surgeon will use ultrasound (US) guidance to locate tumor location during the laparoscopic procedure. The images collected during this process will be recorded by Pathfinder.

DETAILED DESCRIPTION:
The Pathfinder System used during this study is used for data collection purposes only and is not used during the surgical procedure as an image guided system.

Preoperative computed tomography (CT) scans, obtained as standard of care, will be used to generate the image guided liver system 3D liver surface images used during the study.

During the laparoscopic procedure, the Pathfinder device will be inserted through the standard laparoscopic ports (5mm or 10mm) being used for the staging procedure.

A total study population will include 30 subjects: 10 in Phase I and 20 in Phase II that complete the laparoscopic procedure scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for laparoscopic liver ablation procedure
* Had a preoperative CT image that includes the liver

Exclusion Criteria:

* Severe cirrhosis of the liver
* Kidney failure or dialysis
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any subject scheduled for a laparoscopic procedure where liver surface visualization and surface swabbing is feasible with standard port placement.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Phase I: The number of accurate liver surface registrations obtained in the laparoscopic environment providing the surgeon with a comfort level of adding the registration procedure to the scheduled laparoscopic surgical ablation procedure. | 30 days
  Subjects are followed for the study 30days (+/- 14 days) and are considered to have completed the study following this 30 day follow-up visit.
  The performance of accurate physical-to-image registrations obtained during laparoscopic procedures will be evaluated and accepted by the surgeon during the procedure.
Phase II: The number of surgical oblation procedures that present data showing equivalent location of the ablation probe when compared to the US and Pathfinder Guidance System 3D image data. | 30 Days
  The correlation of location of the ablation probe will be evaluated comparing data obtained from the interoperative US images and the data collected with the Pathfinder image guided system.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hansen, M.D., Principal Investigator — PPMC, Liver Cancer Center
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

REFERENCES:
- See also: Pathfinder Company Link — http://www.liversurgery.com